CLINICAL TRIAL: NCT06417632
Title: Prosthetic Outcomes and Clinical Performance of Two Types of Monolithic Zirconia-based Screw-retained Crowns. A Randomized Clinical Trial
Brief Title: Prosthetic Outcomes and Clinical Performance of Implant Supported Zirconia Crowns
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Susan Hattar, Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Susan Hattar
Record Dates: First submitted 2024-01-21; First posted 2024-05-16 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Dental Restoration; Dental Implant
Keywords: implant-supported; patient-reported outcome,; technical, biological outcomes; survival/success rate; single-tooth restorations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graded monolithic Zirconia Crowns (Experimental): 3Y-TZP/5Y-TZP zirconia crown
  Interventions: Other: Graded Zirconia Crown
- Conventional monolithic Zirconia Crowns (Active Comparator): 3Y-TZP zirconia crowns
  Interventions: Other: Conventional Zirconia Crown

INTERVENTIONS:
Other: Graded Zirconia Crown — monolithic implant supported crown
  Arms: Graded monolithic Zirconia Crowns
Other: Conventional Zirconia Crown — monolithic implant supported crown
  Arms: Conventional monolithic Zirconia Crowns

SUMMARY:
To compare biological, technical, radiographic, and patient-reported outcomes of two types of monolithic zirconia crowns screw-retained to implant.

To assess whether the new form of multilayered zirconia crowns will show similar survival and success rate to conventional monolithic Zirconia screw-retained to implants in molar and premolar regions.

First Null Hypothesis: Multilayered monolithic zirconia crowns would have similar survival, success rate compared to conventional monolithic zirconia implant supported crowns.

Second Null hypothesis: There would be no difference in clinical and patients related outcomes between multilayered and conventional monolithic zirconia implant supported crowns.

DETAILED DESCRIPTION:
Study design:

A short-randomized controlled trial study, the (PICO) study design: population will be patients from Jordan University Hospital with implants planned for single screw-retained zirconia crowns in the posterior site (premolar or molar), intervention will be the multilayer monolithic screw-retained zirconia crowns over implants, the comparator is the conventional monolithic zirconia crowns over implants, and the main outcomes will be the prosthetic/technical outcomes, survival and success rates in addition to radiographic, patient-reported outcomes, and biological parameters.

Methodology The patients who fulfilled the inclusion/exclusion criteria and entered the study will have a fully digital workflow starting from data acquisition using an intraoral scanner (3Shape TRIOS® 5) , Ti-base abutment design and CAD/CAM milling of the two types of monolithic zirconia blanks (IPS e.max® ZirCAD Prime and IPS e.max® ZirCAD LT).

The fabricated zirconia crowns in both groups will have the same treatment and will be cemented to the Ti-base abutment according to the (APC) concept; alumina airborne-particle abrasion 50-μm at 1 bar for 15-20 seconds, intaglio surface primed using MDP for 60 seconds and air blown for 5 seconds, and finally cemented to the abutment by phosphate monomer resin cement PANAVIA™ V5(Blatz-Alvarez-Compendium-APC-2016, n.d.).

On the other hand, the Ti-base abutment: height will be standardized at 4mm, and the base abutment surface will have blasting with alumina particles of 50 μm at 2-bar pressure for 15-20 seconds at a 10-mm step-over distance at an angle of 45 degrees.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous area with suitable restorative space more than 5.5 mm
* At least 18 years of age
* Opposing natural teeth or fixed restorations supported by teeth or implants.
* Generally good health (ASA I, ASA II)
* Participant complies with good oral hygiene practices (BOP and PI less than 20%)
* Healthy integrated implant/s without signs of periimplantitis in the posterior site planned for single tooth replacement (in premolar or molar areas)
* Patients received bone-level implants, RC Straumann Implants.

Exclusion Criteria:

* Inability to provide consent.
* Temporomandibular disorders
* Smoking of more than 10 cigarettes per day
* Untreated caries or periodontal disease of remaining dentition

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Technical & Biological Outcomes | Baseline, 6 months, 12 months
  The abutments and restoration will be evaluated clinically by two blinded investigators, according to the modified United States Public Health Service (USPHS) criteria USPHS criteria involve four Scales: Alpha, Bravo, Charlie, Delta The criteria of evaluation include: Restoration fracture, Abutment Fracture, Loosening of the restoration, Screw-access hole restoration, Occlusal Wear, Anatomical Form, Color match, Proximal contact, Occlusal Contact, Marginal Fit, Periodontal parameters.
Survival and Success rate | 6 months, 12 months
  All patients will be evaluated for success and survival of restorations at 6 months and 1 year after placement of the restorations (Follow-ups).
  The success rate is defined as the number of restorations that did not change over time. The survival rate is defined as the number of restorations that did not require replacement.
Patient reported outcomes | 6 months, 12 months
  Patient satisfaction in terms of the shape and shade of the crown, their ability to chew (function) and floss (proximal contact) and their overall satisfaction with the restoration provided will be assessed by a questionnaire based on a five-grade ordinal category scale (extremely satisfied, satisfied, neutral, dissatisfied and extremely dissatisfied). Each patient was asked to fill out the questionnaire themselves to ensure as little bias as possible.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hattar, Professor, Principal Investigator — University of Jordan
Locations (1):
- The university ofJordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le M, Dirawi W, Papia E, Larsson C. Clinical Outcome of Three Different Types of Posterior All-Ceramic Crowns. A 3-Year Follow-up of a Multicenter, Randomized, Controlled Clinical Trial. Int J Prosthodont. 2023 Nov 1;36(5):546-553. doi: 10.11607/ijp.8016. PMID 36484665
- [Background] Hosseini M, Worsaae N, Gotfredsen K. A 5-year randomized controlled trial comparing zirconia-based versus metal-based implant-supported single-tooth restorations in the premolar region. Clin Oral Implants Res. 2022 Aug;33(8):792-803. doi: 10.1111/clr.13960. Epub 2022 Jun 11. PMID 35633183
- [Background] Jung RE, Zembic A, Pjetursson BE, Zwahlen M, Thoma DS. Systematic review of the survival rate and the incidence of biological, technical, and aesthetic complications of single crowns on implants reported in longitudinal studies with a mean follow-up of 5 years. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:2-21. doi: 10.1111/j.1600-0501.2012.02547.x. PMID 23062124
- [Background] Zhang CN, Zhu Y, Zhang YJ, Jiang YH. Clinical esthetic comparison between monolithic high-translucency multilayer zirconia and traditional veneered zirconia for single implant restoration in maxillary esthetic areas: Prosthetic and patient-centered outcomes. J Dent Sci. 2022 Jul;17(3):1151-1159. doi: 10.1016/j.jds.2022.01.012. Epub 2022 Feb 5. PMID 35784115